CLINICAL TRIAL: NCT07200388
Title: The Role of Emotional Granularity in Enhancing Resilience Among Young and Middle-Aged Colorectal Cancer Survivors: A Mixed-Methods Study
Brief Title: How Emotional Granularity Helps Build Resilience in Young and Middle-Aged Colorectal Cancer Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Second Affiliated Hospital of Soochow University (Other); Kunshan First People's Hospital Affiliated to Jiangsu University (Industry)
Responsible Party: Principal Investigator, Dr Joyce Chung, Associate Professor, The Hong Kong Polytechnic University
Other Study IDs: HSEARS20250802001
Record Dates: First submitted 2025-09-17; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Emotional Granularity; Psychological Resilience; Mixed Methods Research; Young and Middle-Aged Adults; Colorectal Neoplasms; Emotional Regulation
MeSH Terms: conditions — Colorectal Neoplasms; Emotional Regulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young and Middle-Aged CRC Survivors: This single cohort consists of young and middle-aged adult survivors of colorectal cancer. All participants will complete the quantitative survey phase. A subset of participants, purposively sampled based on their survey scores, will then be invited to participate in the qualitative interview phase. There is no intervention administered; this is an observational study examining the relationships between emotional granularity, emotion regulation, and resilience.

SUMMARY:
This study aims to understand how the ability to identify and describe specific emotions (called "emotional granularity") influences coping and adaptation ("resilience") in young and middle-aged colorectal cancer survivors.

The main questions to be answer are:

1. How does emotional granularity help build resilience during cancer recovery?
2. How does emotion regulation contribute to resilience building?
3. What specific emotional needs and challenges do survivors experience?

This is an observational study where no experimental treatments are provided. Participants will complete an online questionnaire about background, emotions, ways of managing emotions, and ability to cope with stress. A subset of participants will then be invited to take part in a private, 30-60 minute interview to share personal experiences and feelings in more detail.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a major global public health concern with rising incidence and mortality rates globally. While advances in treatment have improved survival rates, young and middle-aged survivors face unique and complex challenges, including severe emotional distress, disrupted social networks, work-related economic toxicity and concerns regarding fertility, that necessitate tailored psychosocial interventions. Resilience, defined as a dynamic psychosocial outcome enabling individuals to adapt to adversity, has emerged as a crucial determinant of quality of life among CRC survivors. Adaptive emotion regulation is fundamental to fostering resilience, yet existing emotional interventions have predominantly provided general emotion regulation strategies without addressing patients' proficiency in effectively applying these strategies. Emotional granularity, the ability to differentiate and label subtle emotional experiences, is posited to enhance emotion regulation efficacy.

Therefore, to generate an evidence-based blueprint for emotion-focused psychosocial programs designed to strengthen resilience and enhance quality of life among young and middle-aged colorectal cancer survivors. This sequential mixed-methods investigation aims to clarify how emotional granularity influences resilience through emotion regulation, to explore survivors' emotional needs, and to provide evidence for the future intervention design. The inclusion criteria are (1) young and middle-aged adult patients (18-60 years); (2) patients diagnosed with CRC; (3) patients have completed primary treatments without experiencing a recurrence of CRC; and (4) patients able to use a smartphone and agree to participate in the study. The exclusion criteria are (1) patients who have not been informed of their cancer diagnosis due to family decision to withhold information; and (2) patients suffering from severe conditions that may affect participation or assessment.

A cross-sectional questionnaire will first be employed to examine the mediating role of emotion regulation in the relationship between emotional granularity and resilience after providing informed consent. Measures will include demographic information and the Chinese versions of the Range and Differentiation of Emotional Experience Scale, the Difficulties in Emotion Regulation Scale and the 10-item Connor-Davidson Resilience Scale. A total of 236 participants will be recruited from teaching hospitals of Soochow University and Jiangsu University, Suzhou, Jiangsu province. Mediation analysis will examine whether emotion regulation channels the effect of emotional granularity on resilience. The second phase will involve individual, semi-structured interviews lasting thirty to sixty minutes each, purposively sampling 20-25 participants with high, medium and low scores from the first phase.

ELIGIBILITY:
Inclusion Criteria:

* Young and middle-aged adult patients (age in the range of 18-60 years);
* Patients diagnosed with CRC;
* Patients have completed primary treatments (e.g., surgery, chemotherapy, and/or radiotherapy) without experiencing a recurrence of CRC;
* Patients able to use a smartphone and agree to participate in the study.

Exclusion Criteria:

* Patients who have not been informed of their cancer diagnosis due to family decision to withhold information;
* Patients suffering from severe conditions that may affect participation or assessment, such as significant cognitive impairment, psychiatric disorders, or communication disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of samples and data obtained from three major regional tertiary hospitals in Suzhou, Jiangsu Province:
  1. The First Affiliated Hospital of Soochow University: A leading comprehensive tertiary Grade A hospital and a major clinical, teaching, and research center in the region.
  2. The Second Affiliated Hospital of Soochow University: Another key comprehensive tertiary Grade A hospital providing high-level medical services to the urban population.
  3. Kunshan First People's Hospital Affiliated to Jiangsu University: A premier tertiary Grade A hospital representing the high-quality healthcare infrastructure of county-level cities within the Suzhou administrative area.
  This selection encompasses top-tier medical institutions from both the central urban district of Suzhou and a developed county-level city (Kunshan), ensuring a representative and diverse sample of the patient population and healthcare delivery within the Suzhou region.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Level of Resilience | Baseline (Day 1, at questionnaire completion for each participant)
  Resilience will be measured by the total score on the Chinese version of the 10-item Connor-Davidson Resilience Scale (CD-RISC-10). Scores range from 0 to 40, with higher scores indicating higher levels of resilience.

SECONDARY OUTCOMES:
Emotional Granularity Score | Baseline (Day 1, at questionnaire completion for each participant)
  Emotional granularity (the ability to differentiate emotional experiences) will be measured by the total score on the Chinese version of the Range and Differentiation of Emotional Experience Scale (RDEES). The scale contains 11 items, and higher scores indicate a greater ability to differentiate between subtle emotions.
Emotion Regulation Difficulties Score | Baseline (Day 1, at questionnaire completion for each participant)
  Difficulties in emotion regulation will be measured by the total score on the Chinese version of the Difficulties in Emotion Regulation Scale (DERS). The scale contains 36 items, and higher scores indicate greater problems with emotion regulation.

OTHER OUTCOMES:
Qualitative Themes on Emotional Needs | Post-questionnaire phase (within approximately 2-6 weeks after baseline, depending on scheduling of interviews)
  Themes and patterns identified through thematic analysis of semi-structured interviews regarding survivors' emotional experiences, needs, and coping strategies.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Kunshan First People's Hospital Affiliated to Jiangsu University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhu, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided
A final decision regarding sharing individual participant data (IPD) has not yet been finalized. This is due to the need for further internal discussions and consultations with all collaborating institutions, particularly regarding compliance with cross-border data transfer regulations under China's Personal Information Protection Law (PIPL) and ethical guidelines governing participant privacy. Additionally, the feasibility of robust de-identification processes and secure data-sharing mechanisms is being evaluated to ensure participant confidentiality. The final decision will be determined before study completion and will align with journal requirements, participant consent agreements, and institutional policies.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT07200388/Prot_SAP_000.pdf